CLINICAL TRIAL: NCT06326619
Title: Survival Benefit of Palliative Primary Tumor Resection and Systemic Therapy Versus Systemic Therapy Only Among Patients With Stage IV Colorectal Carcinoma
Brief Title: Survival Benefit of Primary Tumour Resection Compared to Systemic Therapy Alone in Stage IV Colorectal Cancer Patients
Acronym: SurvSysT
Status: Completed | Type: Observational
Sponsor: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Collaborators: Clinical-Epidemiological Cancer Registry Brandenburg-Berlin (Unknown)
Responsible Party: Principal Investigator, Rene Mantke, Head of Surgery, Medizinische Hochschule Brandenburg Theodor Fontane
Other Study IDs: SurvSysT
Record Dates: First submitted 2024-03-17; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; Neoadjuvant Systemic Therapy
Keywords: Survival Analysis; Palliative Care; Primary Tumor Resection
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SYST: Systemic treatment only. Systemic treatment was defined as the application of chemotherapy, antibody, or immunotherapy (alone or in combination) starting within 12 months after diagnosis (definition for both groups)
  Interventions: Procedure: Systemic Therapy
- PTR+SYST: primary tumor resection and systemic treatment At least one of the following surgical procedures were performed: German procedure codes OPS 5-455.*, 5-456.*, 5-484.*, 5-485.*
  Interventions: Procedure: Primary tumor resection; Procedure: Systemic Therapy

INTERVENTIONS:
Procedure: Primary tumor resection — In addition to systemic therapy a primary tumor resection was performed.
  Groups: PTR+SYST
Procedure: Systemic Therapy — chemotherapy, antibody, or immunotherapy (alone or in combination) starting within 12 months after diagnosis

SUMMARY:
About 20-25 percent of all colorectal cancer patients are diagnosed with International Union Against Cancer (UICC) stage IV disease. The benefit of primary tumor resection in the palliative context is therefore of high concern. However, empirical evidence from randomized and observational studies is inconsistent.

The objective of the present study is to compare the survival of palliative stage IV colorectal cancer patients selected for primary tumor resection and systemic treatment (PTR+SYST) to patients with systemic treatment only (SYST).

DETAILED DESCRIPTION:
Mortality after PTR+SYST compared to SYST alone was evaluated in a retrospective observational cohort of patients diagnosed from 2012-2020 in the cancer registry in the federal state of Brandenburg (Germany), excluding patients with rectal cancer of the lower two-thirds, emergency procedures, unknown Eastern Cooperative Oncology Group Score (ECOG) status, ECOG>2, unknown metastatic status or unclear grading.

PTR was defined as resection of the primary tumor within 12 months after diagnosis (German procedure codes [Operationen- und Prozedurencodes, OPS] 5-455.*, 5-456.*, 5-484.*, 5-485.*). Cases with additional, but incomplete, resection of metastases were included. SYST was defined as the application of chemotherapy, antibody, or immunotherapy (alone or in combination) starting within 12 months after diagnosis.

The primary study endpoint was mortality. Survival of treatment groups (PTR+SYST vs. SYST) was compared using Kaplan-Meier survival plots and log-rank tests. Follow-up started at diagnosis and ended at death or December 31, 2020, whichever came first. Hazard ratios (HR) were calculated with multivariate Cox regression adjusting for sex (male, female), age at diagnosis (in years), ECOG status (0, 1, 2), localization and number of metastases according to TNM, 8th edition (M1a, M1b, M1c), grading (G1-2, G3-4), and localization of the primary tumor (colon carcinoma on the right side, colon carcinoma on the left side, or rectum carcinoma upper third).

Sensitivity analyses were performed to reduce indication bias. Propensity score matching was conducted based on a propensity score determined by logistic regression of treatment (PTR+SYST vs. SYST) on the same variables as above plus radiotherapy (yes/no). For each patient in the SYST group, a patient from the PTR+SYST group was randomly chosen with the same propensity score as the SYST patient, within a certain margin. The same analyses as above were performed on the matched patient groups. Delayed entry was used to account for the fact that patients who underwent PTR must survive from the date of diagnosis to the date of surgery to be included in the PTR+SYST group, whereas no such requirement was made for patients in the SYST group. Follow-ups started 3, 6, 9, and 12 months after diagnosis, excluding patients who died prior to this time irrespective of treatment (according to the "landmark" approach, as described by Alawadi et al., 2017).

Registry quality assurance measures and procedures:

Quality of German Clinical Cancer Registries have been analysed and described in detail by various publications (for example, PubMed-ID (PMID): 37568750; PMID: 28639952; PMID: 26474650; PMID: 25523845). In summary, the completeness and quality of the data can be rated as high to very high. The basis for this are the statutory reporting requirements, a high reporting fee by European standards for both the registries and the transmitting agent, regular quality conferences, highly standardised documentation requirements for the data transmission, specifications on register-related quality indicators (e.g. completeness), internal data validation measures and a secure and independent funding basis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed colorectal carcinoma
* stage IV
* systemic therapy, starting within 12 months after diagnosis

Exclusion Criteria:

* rectal cancer of the lower two-thirds
* emergency procedures
* unknown Eastern Cooperative Oncology Group (ECOG) performance status
* ECOG>2
* unknown metastatic status
* unclear grading

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Complete residential population of the federal states Brandenburg and Berlin, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Survival | 5-year follow up
  No mortality; no death by any cause; overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Rene Mantke, M.D., Principal Investigator — Medizinische Hochschule Brandenburg CAMPUS GmbH

IPD SHARING:
Plan to Share IPD: No
Individual patient data is not available.

REFERENCES:
- [Derived] Mantke R, Schneider C, von Ruesten A, Hauptmann M. Patients with stage IV colorectal carcinoma selected for palliative primary tumor resection and systemic therapy survive longer compared with systemic therapy alone: a retrospective comparative cohort study. Int J Surg. 2024 Oct 1;110(10):6493-6500. doi: 10.1097/JS9.0000000000001838. PMID 38935125